CLINICAL TRIAL: NCT02444468
Title: A Randomized Study of In-cast Intermittent Pneumatic Foot-compression in the Preoperative Treatment of Malleolar Fractures
Brief Title: Preoperative Treatment of Malleolar Fractures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital of Southern Jutland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IPC-study
Record Dates: First submitted 2015-04-28; First posted 2015-05-14 (Estimated); Last update posted 2016-08-18 (Estimated); Status verified 2016-08

CONDITIONS: Ankle Fractures; Intermittent Pneumatic Compression; Comparative Study; Preoperative Care
MeSH Terms: conditions — Ankle Fractures | interventions — Bandages

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IPC and bandage (Experimental): Pneumatic device and bandage
  Interventions: Device: Flowtron ACS800; Other: Bandage
- Bandage only (Active Comparator): Bandage only
  Interventions: Other: Bandage

INTERVENTIONS:
Device: Flowtron ACS800 — Flowtron ACS800 and bandage
  Arms: IPC and bandage
Other: Bandage — Bandage only

SUMMARY:
This study investigates, in a randomized setting, the use of intermittent in-cast pneumatic foot-compression (IPC) in the preoperative treatment of malleolar fractures. This is to investigate whether the IPC has any effect on preventing swelling of the ankle, and thereby preventing delay of surgery due to swelling.

The investigators will include patients with malleolar fractures that require surgery in two groups, IPC and bandage or bandage only, and measure the time from diagnosis-to-surgery.

DETAILED DESCRIPTION:
Malleolar fractures are often complicated by tissue swelling due to soft tissue injury, haemorrhage and secondary inflammation.

This can lead to severe oedema which can compromise the ability to perform surgery due to blister formation or the inability to close the skin after surgery. Studies have shown that the use of intermittent pneumatic foot-compression (IPC) can reduce waiting time from diagnosis to surgery as well as reduce length of hospital stay.

Purpose of the study is in a randomized study to investigate whether patients requiring surgery because of malleolar fractures has a lower diagnosis-to-surgery time when using IPC than patients not using IPC.

All patients age 18 or above admitted to our hospital with malleolar fractures (AO type 44-A, 44-B, 44-C) requiring surgery, will be randomized to either in-cast IPC or only cast-immobilization. Time from diagnosis of the fracture(time of the x-ray) until start of surgery(time of incision) will be the primary outcome. Patients will be seen in a postoperative ambulatory follow-up at 14 days, 6 weeks, 3 months and 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Malleolar fracture requiring surgery.

Exclusion Criteria:

* Severe arteriosclerosis.
* Known or suspected acute DVT or flebit.
* Severe decompensated heart failure.
* Pulmonary embolism.
* Acute skin conditions as dermatitis, infected wounds or recent skintransplant.
* Open fracture.
* Inability and/or unable to comply with treatment regime and/or to attend postoperative ambulatory follow-up.
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2015-03; Primary Completion 2017-04 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Time from diagnosis-to-surgery | 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Jesper O Schønnemann, Dr, Principal Investigator — Hospital southern Jutland
Locations (1):
- Jesper O. Schønnemann, Aabenraa, Denmark